CLINICAL TRIAL: NCT00200330
Title: Modifying Obesogenic Homes: Impact on Weight Maintenance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HL077082 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2005-09

CONDITIONS: Obesity
Keywords: weight loss; physical activity; diet; home environment
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

INTERVENTIONS:
Behavioral: Behavioral weight loss treatment
Behavioral: Behavioral and home environment weight loss treatment

SUMMARY:
The obesity epidemic observed in recent years can be largely attributed to an obesogenic environment that encourages overeating and sedentary lifestyles. Behavioral weight control treatment, the most empirically validated intervention approach, produces initial weight losses of 10%; however, maintenance of initial weight loss and behavior change has not been achieved. These disappointing long-term results may reflect the fact that participants are given only minimal, indirect instruction on how to change their environment to support their new weight-regulating behaviors. While in theory, the behavioral model emphasizes environmental antecedents and consequences of eating and exercise, in practice, only 1 to 2 sessions in standard treatment are dedicated to stimulus control-types of skills. By teaching weight control skills in a contextual vacuum, participants remain vulnerable to the same environmental influences that maintained their unhealthy eating and exercise habits. Given that the majority of eating and exercise is home-based, a logical step in strengthening behavioral treatment and moving toward an ecological model of behavior is to expand the focus of treatment from the individual to the individual plus their home environment. We propose to test the long-term impact of a behavioral weight control program designed to directly modify both the physical and social home environment of weight loss participants. Two hundred overweight and obese men and women will be randomly assigned to either 18 months of standard behavioral treatment (SBT) or 18 months of standard behavioral treatment plus direct modifications to the home environment (SBT+Home). SBT+Home will incorporate many strategies that have shown promise in improving weight loss (e.g., food and exercise equipment provision, spouse involvement) but will be the first to study both physical and social factors within the home simultaneously and will be the longest examination of the home environment conducted to date. Participants and spouses will be assessed at baseline, 6, 12, and 18 months. We hypothesize that by broadening the focus of treatment from the individual to the individual plus their home environment, SBT+Home will produce both better long-term weight loss and better maintenance of initial weight loss and behavior change. This home environmental approach, if successful, has potential applications to the maintenance of other important health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* are between 21-70 years of age.
* have a body mass index (BMI) between 25-50 kg/m2 .
* live with another overweight adult who is between 18-70 years of age and has a BMI between 25-50 kg/m2 and who is willing to participate in the study

Exclusion Criteria:

* report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q; items 1-4). Individuals endorsing joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
* report conditions that in the judgment of the Principal Investigator would render them potentially unlikely to follow the protocol for 18 months including an illness likely to be terminal within 18 months, plans to move out of the area, substance abuse or other significant psychiatric problems, or dementia.
* report being unable to walk 2 blocks (1/4 mile) without stopping.
* are currently participating in a weight loss program and/or taking a weight loss medication.
* are currently pregnant or intend to become pregnant in the next 18 months.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-11; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Weight loss

SECONDARY OUTCOMES:
Diet composition
Physical activity
Changes in home environment

CONTACTS AND LOCATIONS:
Overall Officials: Amy Gorin, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center, The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Cornelius T, Gettens K, Gorin AA. Dyadic Dynamics in a Randomized Weight Loss Intervention. Ann Behav Med. 2016 Aug;50(4):506-15. doi: 10.1007/s12160-016-9778-8. PMID 26865258
- [Derived] Gorin AA, Powers TA, Koestner R, Wing RR, Raynor HA. Autonomy support, self-regulation, and weight loss. Health Psychol. 2014 Apr;33(4):332-9. doi: 10.1037/a0032586. Epub 2013 Jun 3. PMID 23730718
- [Derived] Gorin AA, Raynor HA, Fava J, Maguire K, Robichaud E, Trautvetter J, Crane M, Wing RR. Randomized controlled trial of a comprehensive home environment-focused weight-loss program for adults. Health Psychol. 2013 Feb;32(2):128-37. doi: 10.1037/a0026959. Epub 2012 Feb 6. PMID 22309885
- See also: Provides description of ongoing studies at the Weight Control and Diabetes Research Center — http://weightresearch.org